CLINICAL TRIAL: NCT05049421
Title: Right Ventricular Function After Coronary Artery Bypass Grafting The SWEDEGRAFT Right-Heart-Substudy
Brief Title: The SWEDEGRAFT Right-Heart-Substudy
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Ivy susanne Modrau, MD, Consultant Cardiac Surgeon, Associate Professor, Aarhus University Hospital Skejby
Other Study IDs: 1-10-72-207-18-2
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Coronary Artery Bypass Surgery; Right-Sided Heart Failure
Keywords: 2-D Echocardiography; 3-D Echocardiography; Coronary Artery Bypass Surgery; Right-Sided Heart Failure; Patient Reported Outcome Measures
MeSH Terms: conditions — Heart Failure | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients following CABG: Recruitment amongst patients enrolled in SWEDEGRAFT RCT at Aarhus University Hospital scheduled for follow-up
  Interventions: Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Echocardiography — Full 2D and 3D echocardiography with special focus on right ventricular function

SUMMARY:
BACKGROUND

Right ventricular dysfunction is a common echocardiographic finding after cardiac surgery. Pericardial disruption has been suggested as the most probable cause as the phenomenon occurs within minutes after pericardial incision.

The investigators suspect that validated two-dimensional echocardiographic measures for right ventricular function might not reflect the altered RV contraction pattern including paradoxical interventricular septal motion and reduced long-axis function following open cardiac surgery.

The present study aims to determine the prevalence and scale of right ventricular dysfunction two years after CABG by applying the latest available two- and three-dimensional echocardiographic technology in right ventricular evaluation. In addition, the investigators investigate the impact of right ventricular dysfunction on functional outcome.

METHODS

The Right-Heart-Study is an observational substudy of the SWEDEGRAFT trial at Aarhus University Hospital in Denmark. SWEDEGRAFT is a nordic, multicenter, prospective, randomized, register-based, clinical trial (ClinicalTrials.gov Identifier: NCT03501303; Ragnarsson 2020). Patients for the current Right-Heart-Substudy will be recruited amongst the 269 patients included in the SWEDEGRAFT trial at Aarhus University Hospital from 10 September 2018 to 25 May 2020. Patients are enrolled at the time of SWEDEGRAFT follow-up with cardiac-CT (approximately 30 months after CABG). After written informed consent, we perform additional full 2D and 3D echocardiography with special focus on RV function, collect patient-reported data on functional outcome, and measure brain natriuretic peptide and hemoglobin levels.

DETAILED DESCRIPTION:
Complete study protocol attached

ELIGIBILITY:
Inclusion Criteria:

SWEDEGRAFT inclusion criteria:

* First-time non-emergent CABG patients
* Need for at least one vein graft
* Able to provide informed consent and accepted for isolated primary CABG.

Additional inclusion criteria for the Right-Heart-Substudy:

• Ability to meet for follow-up visit

Exclusion Criteria:

SWEDEGRAFT exclusion criteria:

* No greater saphenous vein grafts available (previous vein stripping or poor vein quality)
* Age > 80 years at the time of inclusion
* Allergy to contrast dye
* Renal failure with eGFR <15 ml/min at primary inclusion
* Coagulation disorders
* Excessive risk of wound infection
* Participation in other interventional trial on grafts
* Any condition that seriously increases the risk of non-compliance or loss of follow-up
* Pregnant women or women of child bearing potential without negative pregnancy test

Additional inclusion criteria for the Right-Heart-Substudy:

• Inability to cooperate to transthoracic echocardiography

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients enrolled in the SWEDEGRAFT RCT due to 2,5 year follow-up. Patients have undergone elective stand-alone first-time coronary artery bypass grafting
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
3D right ventricular ejection fraction | 30 months postoperative
  Right ventricular function assessed by 3D echocardiography
Right ventricular strain | 30 months postoperative
  Derived from two-dimensional speckle-tracking

SECONDARY OUTCOMES:
Disease-specific health-related quality of life | 30 months postoperative
  Seattle Angina Questionnaire-7
  -> 0 denotes the worst and 100 the best possible health status
Degree of dyspnea at exertion | 30 months postoperative
  NYHA class
Perceived exertion during exercise | 30 months postoperative
  Borg CR10® Scale
  -> Range from 0: No exertion to 10: Maximal level of exertion
Pro-Brain Natriuretic Peptide | 30 months postoperative
  pg/mL
Long-term Major Adverse Cardiac and Cerebrovascular Events | 5 and 10 years after CABG
  all-cause mortality, myocardial infarction, repeat hospitalization due to cardiac cause, cerebrovascular accident, repeat revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Ivy Modrau, MD, dr.med., Principal Investigator — Aarhus University Hospital Skejby
Locations (1):
- Aarhus University Hospital Skejby, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ragnarsson S, Janiec M, Modrau IS, Dreifaldt M, Ericsson A, Holmgren A, Hultkvist H, Jeppsson A, Sartipy U, Ternstrom L, Per Vikholm MD, de Souza D, James S, Thelin S. No-touch saphenous vein grafts in coronary artery surgery (SWEDEGRAFT): Rationale and design of a multicenter, prospective, registry-based randomized clinical trial. Am Heart J. 2020 Jun;224:17-24. doi: 10.1016/j.ahj.2020.03.009. Epub 2020 Mar 13. PMID 32272256

DOCUMENTS (1):
  • Study Protocol (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT05049421/Prot_000.pdf